CLINICAL TRIAL: NCT03291964
Title: QuickBrain MRI for Acute Pediatric Head Trauma
Brief Title: Rapid MRI for Acute Pediatric Head Trauma
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dr. David Sheridan, Assistant Professor of Emergency Medicine/Pediatrics, Oregon Health and Science University
Other Study IDs: 17254
Record Dates: First submitted 2017-06-27; First posted 2017-09-25 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Head Trauma; Image, Body
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid Brain MRI — Children undergoing head CT for evaluation of acute head injury will also undergo rapid brain MRI with GRE sequence that is specific for blood. Their clinical care will not change at all based on the MRI.

SUMMARY:
Pediatric head trauma is a leading cause of morbidity and mortality for children/adolescents. The current standard of care regarding imaging modality when concerned for an acute head injury is CT. This exposes children to radiation that may predispose to future malignancy. Rapid MRI is a test that eliminates radiation and has expanded uses in multiple other areas. This study is evaluating it for pediatric acute head trauma.

DETAILED DESCRIPTION:
Initial retrospective study suggests that QbMRI has adequate sensitivity to detect acute ciTBIs in children. This preliminary study included all pediatric trauma patients presenting to OHSU from 2/2010 through 12/2013 who had both a head CT and QbMRI. The current standard of care in the pediatric ICU at OHSU is for patients admitted with an acute head injury to undergo routine QbMRI follow up to assess status of the injury rather than a repeat head CT. Our study team collected clinical data on these patients that included clinical interventions and then de-identified all head CT and QbMRI images for this cohort. The images were then independently reviewed by 2 neuroradiology fellows at OHSU (Please refer to Figure 1). The sensitivity of QbMRI to detect any radiographic injury was 85% (95% CI: 73, 93), but increased when evaluating clinically important TBIs to 100% (95% CI: 89, 100). The largest limitation of this study was the variable and often long time interval between acquisition of the head CT and QbMRI. The average length of time between the initial head CT and QbMRI was 27.5 hours with only 41% receiving both imaging tests within 12 hours of each other. Also, preliminary data was collected by retrospective review. As such, it is very promising that initial study had high sensitivity, but further prospective pilot data with a shorter interval between the index and reference test is needed to assess the discrepancy between the two types of lesions (radiographic vs clinically important) and feasibility of obtaining qbMRI in the setting of acute pediatric head trauma. While this study did not miss any clinically important TBIs, on further review of radiographic "missed lesions", the study pediatric neurosurgeon noted signs of a healing bleed. This may suggest that they were "missed" because they were healed rather than present and not seen. All patients that did not have a lesion identified on QbMRI did not require significant clinical interventions and only underwent periods of observation in the hospital. However, this raises the need for a prospective trial to obtain QbMRI imaging within the same time frame sequentially after the initial head CT.

ELIGIBILITY:
Inclusion Criteria:

1. The patient presents to the pediatric emergency department or trauma system at OHSU or is a trauma system transfer patient to OHSU
2. Age 0-14 years.
3. Being evaluated for a traumatic head injury and attending physician decides to obtain a head CT.
4. Clinically stable for additional testing: provider deems it safe to obtain a QbMRI in the ED without deep sedation

Exclusion Criteria:

1. Subject is from outside hospital and head CT was performed greater than 6 hours prior
2. Subject is from outside hospital and initial head CT is not in our imaging system for review
3. History of intracranial surgery
4. History of metallic implants making MRI contraindicated
5. Decompressive surgery prior to QbMRI

Ages: 0 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: All pediatric trauma patients being evaluated with a head CT for acute intracranial injury
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-09-03 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sheridan, MD MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Quick Brain: Pediatric head trauma patients
Period: Overall Study
Arm/Group | Quick Brain
Started | 73
Completed | 73
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: children being evaluated in the ED for head trauma.
Arm/Group | Quick Brain
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 73
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 4.0 [1 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 73
Region of Enrollment [Number; unit: participants]
  United States | 73

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity: Percentage of MRIs Correctly Identifying Clinically Important Intracranial Injury (True Positives)
Description: Sensitivity of Rapid MRI for detection of a clinically important intracranial injury: Percentage of MRIs identifying clinically important intracranial injury. Sensitivity was calculated as the number of true positives divided by "true positive plus false negative". True positive was defined based on meeting clinical criteria for a clinically important TBI and if the imaging found the injury.
Time Frame: within 6 hours from the initial head CT
Measure: Number; unit: Percentage of MRIs correctly identifying
Arm/Group | Quick Brain
Number analyzed (Participants) | 73
Percentage of MRIs correctly identifying | 70

2. Secondary Outcome: Time From Order to Obtaining MRI
Description: minutes
Time Frame: During initial ER stay within 3 hours from time of entry to the ER
Reporting Status: Not Posted

3. Secondary Outcome: Need for Anxiolysis Medication (Defined as Benzodiazepines for Imaging Indication)
Description: Number of patients requiring medication to obtain imaging
Time Frame: During initial ER stay within 3 hours from time of entry to the ER
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Quick Brain
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03291964/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03291964/ICF_001.pdf